CLINICAL TRIAL: NCT06621719
Title: Evaluation of Secondary Alveolar Cleft Reconstruction Using Bone Matrix Prepared From Cancellous Particulates Mixed With Albumin-PRF or L-PRF: (A Randomized Controlled Clinical Trial)
Brief Title: Evaluation of Secondary Alveolar Cleft Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ahmed Nagi Alghandour, Lecturer, Beni-Suef University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23
Record Dates: First submitted 2024-09-29; First posted 2024-10-01 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Alveolar Cleft

STUDY DESIGN:
Intervention Model Description: This clinical trial introduces a radiographic volumetric and bone density comparison of alveolar clefts obliterated with "sticky bone," prepared by mixing iliac crest cancellous bone particulates with either L-PRF (Control group) or Albumin-PRF (Study group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (L-PRF) (Active Comparator): The tubes will be centrifuged at (700 g for 12 min). By the end of the centrifuge cycle, the PRF clots will be extruded from the tubes with a sterile tweezer and separated from the underlying RBCs with sterile scissors.
  Interventions: Procedure: Alveolar Cleft Reconstruction
- Study group (Albumin-PRF) (Active Comparator): The tubes will be centrifuged at (700 g for 8 minutes). The upper (PPR) layer will be aspirated through the unremoved plastic cap, collected in a 2-ml plastic syringe, and placed into a bio-heat device for heating at (75°C for 10 minutes) for the purpose of albumin gel formation, which will be allowed to cool for an additional ten minutes into the room temperature in a sealed dark container before being mixed with the liquid PRF and buffy coat lower layers, using a female-female luer lock connector
  Interventions: Procedure: Alveolar Cleft Reconstruction

INTERVENTIONS:
Procedure: Alveolar Cleft Reconstruction — Alveolar Cleft Reconstruction Using Bone Matrix Prepared from Cancellous Particulates Mixed with Albumin-PRF in study group versus L-PRF in control group

SUMMARY:
The rehabilitation of the disorganized maxilla is the primary objective of secondary alveolar bone grafting (SABG) for alveolar clefts, as the bony reconstruction of the discontinued maxillary arch would permit proper anterior teeth eruption, improve their orthodontic movements, restore the nasal and alar base symmetry, counteract the growth disturbance effects and seal the oronasal communication. By the time the transverse growth of the maxillary arch is nearly complete during the mixed dentition stage, (SABG) intends to bridge the maxillary continuity by a quantitative bone graft entity that minimizes the maxillary collapse and growth impairment after an appropriate separation and elevation of the nasal and mucosal flaps.

DETAILED DESCRIPTION:
By its ample content of subcutaneous autogenous cancellous bone particulates, the iliac crest is considered the gold standard for (SABG) of alveolar clefts, with optimal restoration of the maxillary continuity, and fair subsequent teeth eruption, orthodontic movements or implant placement. However, several studies have demonstrated that the final volume of the sole iliac crest particulate graft is unpredictable.

Sohn et al. in 2010 introduced the growth-factors enriched bone matrix "sticky bone" concept that incorporates the platelet-rich fibrin (PRF) into the particulate grafts to enhance their moldability and enrich them with three-dimensional (3D) fibrin networking scaffold and high concentrations of growth factors, which promote cell division, modulate tissue healing and induce angiogenesis, such as vascular endothelial growth factors (VEGF), recombinant human platelet-derived growth factor (rhPDGF), transforming growth factors ß-1 (TGFß-1), bone morphogenic protein-2 (rhBMP2), insulin growth factor-I (IFG-I), and epithelial growth factor (EGF), and interleukins.

During the last decade, various (PRF) preparations and centrifuge protocols have been developed, forming various platelet products with different biological constitutions and potential applications. The (PRF) evolution began with the development of the leukocyte- and platelet-rich fibrin (L-PRF) by an increased centrifuge time and speed, followed by advanced platelet-rich fibrin (A-PRF), injectable platelet-rich fibrin (I-PRF), horizontal platelet-rich fibrin (H-PRF), Concentrated PRF (C-PRF) and most recently the albumin-PRF (Albumin gel).

The (L-PRF) employs the extract of the platelet-rich plasma (PRP) in the form of a fibrin clot, meanwhile discarding the platelet-poor plasma (PPP). On the other hand, the albumin gel preparation employs the aspiration and heating of the platelet-poor plasma (PPP), the upper layer, then remixing it with the (PRP) layer and the buffy coat; the lower layers, after being allowed to cool. Although the heating and cooling process would threaten the vitality of cells and the growth factor of the (PPP) layer, this will polymerize its plasmatic proteins and denature the high albumin content as a result of the replacement of the weak hydrogen bond linkages within the protein molecule, with densely organized ones, in addition to the formation of thermal aggregate cross-linkage fibrin networks with an overall endured mechanical strength, prolonged degradation time up to 4-6months, and extended release of growth factors up to ten days.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes with unilateral secondary maxillary alveolar cleft, during the mixed dentition stage with an age range of (eight to twelve years old)
2. Good general good health and proper state of oral hygiene.

Exclusion Criteria:

1. The detection of maxillary pathosis or palatal fistulae during the radiographic or clinical examination.
2. Patients with systemic disorders that would compromise the bone harvest or graft outcomes, those with cleft-associated syndromes or a history of previous failed (SABG)

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
The graft fill rate | 6 months
  The patients will be followed up immediately after surgery and then monthly during the six-month graft consolidation period.
  Immediate postoperative and six-month postoperative Cone beam xray will be undertaken for the patients, which will be superimposed to compare the exact extent of vertical and horizontal bone loss between the cases of the study and control groups.
The graft resorption rate | 6 months
  The patients will be followed up immediately after surgery and then monthly during the six-month graft consolidation period.
  Immediate postoperative and six-month postoperative Cone beam xray will be undertaken for the patients, which will be superimposed to compare the exact extent of vertical and horizontal bone loss between the cases of the study and control groups.
The bone bridge formation rate | 6 months
  The patients will be followed up immediately after surgery and then monthly during the six-month graft consolidation period.
  Immediate postoperative and six-month postoperative Cone beam xray will be undertaken for the patients, which will be superimposed to compare the exact extent of vertical and horizontal bone loss between the cases of the study and control groups.
Bone bridge density values: | 6 months
  The patients will be followed up immediately after surgery and then monthly during the six-month graft consolidation period.
  Immediate postoperative and six-month postoperative Cone beam xray will be undertaken for the patients, which will be superimposed to compare the exact extent of vertical and horizontal bone loss between the cases of the study and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef University, Giza, Cairo Governorate, Egypt